CLINICAL TRIAL: NCT07238205
Title: The Effect of Mixed Reality Application in Teaching Cervical Effacement and Dilatation on Cognitive Load, Sense of Presence, and Midwifery Professional Perception
Brief Title: Mixed Reality Training for Teaching Cervical Effacement and Dilation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Ulkin Gündüz, Research Assistant, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MAU-Midwifery-UG-01
Record Dates: First submitted 2025-09-12; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Labor; Poor, Primary
Keywords: Cervical Dilatation; Labor; First Stage

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group controlled trial including an intervention group receiving mixed reality training and a control group receiving standard education.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded to group allocation, and the outcomes assessor was blinded to the intervention received by each participant to prevent assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed Reality Training Group (Experimental): Students will participate in a mixed reality (MR)-based training program.
  Interventions: Other: mixed reality education
- Standard Education Group (Active Comparator): Students in the control group will receive traditional theoretical instruction.
  Interventions: Other: Standard Education Group

INTERVENTIONS:
Other: mixed reality education — Students will participate in a mixed reality (MR)-based training program.
  The program is designed to teach cervical effacement and dilation assessment.
  During the training, students will interact with three-dimensional virtual cervical models.
  They will be able to practice repeatedly in a safe, error-free environment to enhance their clinical skills.
  After completing MR training, students will perform vaginal examinations on 10 virtual patient scenarios.
  The accuracy of each assessment will be automatically evaluated by the system.
  Following MR training, students will conduct vaginal examinations on five pregnant women under researcher supervision in a real clinical setting.
  The following scales will be administered to participants:
  Cognitive Load Scale
  Sense of Presence Scale
  Midwifery Professional Perception Scale
  These measures will be used to determine the cognitive and professional effects of MR-based learning.
  Arms: Mixed Reality Training Group
Other: Standard Education Group — Students in the control group will receive traditional theoretical instruction.
  The training content will cover the principles of cervical effacement and dilation assessment.
  After completing the theoretical training, students will complete the Cognitive Load Scale and the Midwifery Professional Perception Scale.
  Under researcher supervision, students will perform vaginal examinations on five pregnant women to assess cervical effacement and dilation.
  These evaluations will be used to examine the effects of traditional training on students' cognitive load, professional perception, and practical assessment skills.
  Arms: Standard Education Group

SUMMARY:
The aim of this educational research is to determine whether a mixed reality-based training program is effective in teaching midwifery students how to assess cervical effacement and dilation. The study also examines the impact of mixed reality on students' cognitive load, sense of presence, and midwifery professional perception.

The main questions the study seeks to answer are:

Does mixed reality training reduce students' cognitive load?

Does mixed reality increase the students' sense of presence?

How does mixed reality-based training influence students' professional perception of midwifery?

Do students who receive mixed reality training perform better in assessing cervical effacement and dilation on real pregnant women compared with the control group?

DETAILED DESCRIPTION:
The aim of this educational research is to determine whether a mixed reality-based training program is effective in teaching midwifery students how to assess cervical effacement and dilation. The study also examines the impact of mixed reality on students' cognitive load, sense of presence, and midwifery professional perception.

The main questions the study seeks to answer are:

Does mixed reality training reduce students' cognitive load?

Does mixed reality increase the students' sense of presence?

How does mixed reality-based training influence students' professional perception of midwifery?

Do students who receive mixed reality training perform better in assessing cervical effacement and dilation on real pregnant women compared with the control group?

How the research will be conducted:

Researchers will compare a mixed reality intervention group with a control group receiving traditional training. Students in both groups will evaluate five different pregnant women to assess cervical effacement and dilation in real clinical settings.

Participants will:

Receive either mixed reality-based training (intervention) or traditional instruction (control)

Complete the Cognitive Load Scale, Sense of Presence Scale, and Midwifery Professional Perception Scale

Perform cervical effacement and dilation assessments on five pregnant women during clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the Midwifery Department at Mardin Artuklu University,
* Taking the course "Normal Birth and Postpartum Care,"
* Who have not previously received any structured training (practical training, simulation, etc.) related to vaginal examination or cervical dilation/effacement procedures,
* Who do not feel confident in assessing cervical effacement and dilation,
* Who volunteer to participate in the study will be included,
* Pregnant women who are in the first stage of labor and have no obstetric complications.

Exclusion Criteria:

* Individuals who are graduates of health vocational high schools,
* Have disabilities in their eyes, hands, arms, or fingers,
* Those who do not complete the training will not be included.

Ages: 18 Months to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Cervical Dilation Measurement (cm) | 4 month
  Accuracy of cervical dilation measurement will be assessed by calculating the absolute difference (in centimeters) between the student's measurement and the researcher's reference measurement. Each participant will perform one vaginal examination on five different pregnant women. The mean absolute difference across all five assessments will be reported as the participant's cervical dilation measurement accuracy. Smaller values indicate higher accuracy.
Accuracy of Cervical Effacement Measurement (%) | 4 month
  Cervical effacement accuracy will be assessed by calculating the absolute difference (in percentage points) between the student's effacement measurement and the researcher's reference measurement. Each participant will perform one vaginal examination on five different pregnant women. The mean absolute difference across all five assessments will be reported as the participant's cervical effacement measurement accuracy. Smaller values indicate higher accuracy.

SECONDARY OUTCOMES:
Assessment of Cognitive Load | 4 months
  Cognitive load will be assessed using the Cognitive Load Scale, a 9-point Likert-type measure.
  Participants will respond to the question "How much mental effort did you invest in completing the task?" by selecting a score between 1 (low) and 9 (high).
  The midpoint of the scale is 5; participants scoring above this value will be considered to have experienced higher levels of cognitive load.
Assessment of Presence Experience | Immediately after MR training (within 1 day)
  The sense of presence will be assessed using the Presence Scale (PS) adapted to a 5-point Likert scale. Participants will rate their virtual reality experience from 1 (strongly disagree) to 5 (strongly agree). Higher subscale scores indicate that the virtual environment is perceived as more realistic and that the sense of presence is stronger.
Assessment of Midwifery Professional Perception | 4 months
  Midwifery professional perception will be assessed using the Midwifery Professional Perception Scale (MPPS). Participants will rate statements reflecting their perceptions of the midwifery profession on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate a more positive perception of the midwifery profession.

CONTACTS AND LOCATIONS:
Overall Officials: Ülkin Gündüz Aruser, Ph.D, Principal Investigator — Mardin Artuklu University; Hacer Ünver Koca, Assoc. Prof., Study Director — Inonu University
Locations (1):
- Mardin Training and Research Hospital, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No